CLINICAL TRIAL: NCT02798796
Title: Brazilian Randomized Study - Impact of Preoperative Magnetic Resonance in the Evaluation for Breast Cancer Conservative Surgery
Brief Title: Brazilian Randomized Study - Impact of MRI for Breast Cancer
Acronym: BREAST-MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 974.504
Record Dates: First submitted 2015-08-03; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; conservative surgery; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI Group (Experimental): MRI Group - all patients will be submitted to clinical examination, mammography and / or ultrasound, and breast MRI
  Interventions: Device: MRI
- Control Group (No Intervention): Control group - all patients will be submitted to clinical examination, mammography and / or ultrasound of the breasts.

INTERVENTIONS:
Device: MRI — All patients will be submitted to MRI
  Arms: MRI Group

SUMMARY:
The aim of this study is to evaluate the ability of MRI to select patients for conservative treatment of breast cancer. Participants: female, over 18 years with breast cancer, stages I, II and III candidates for conservative surgery will be randomly randomized to do MRI or not according mammary density.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the ability of MRI to select patients for conservative treatment of breast cancer.An accurate assessment of the tumor is essential to select the best therapeutic strategy in the treatment of breast cancer.Currently, mammography, ultrasound and clinical examination are the standard techniques to assess the extent and location of the tumor.However, these imaging methods fail to assess the real size in approximately one third of patients eligible to conservative treatment.MRI has high sensitivity (95-100%) in the detection of invasive cancers as well as being able to detect hidden tumors, multifocality, multicentricity and cancer in the contralateral breast more often and greater accuracy than mammography or ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Over 18 years with breast cancer
* Clinical stages I, II and III candidates for conservative surgery

Exclusion Criteria:

* Contra-indication for breast MRI (ex. Metal implant)
* Claustrophobia
* Impossibility to stay in the prone position for more than an hour
* History of allergic reaction to the paramagnetic contrast
* History of chronic kidney disease on dialysis
* Personal history of breast cancer treated surgically in the last 12 months.
* Pregnancy or breastfeeding past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
False positive rate, false negative rate, positive predictive value and negative predictive value MRI in the Breast Cancer conservative surgery | 3 years

SECONDARY OUTCOMES:
Describe the percentage of positive margins on pathological examination | 3 years
Describe the percentage of additional surgery rates | 3 years
Describe the percentage surgical change from conservative surgery to mastectomy | 3 years
Calculate the False positive rate, false negative rate , positive predictive value and negative predictive value according mammographic density, molecular subtype and histopathology of the tumor | 3 years
Calculate the period after successful treatment in which there is no appearance of the symptoms or effects of the disease after 3 and 5 years bettwen groups | 5 years
Calculate how much is the cost to do the exam considering the false positive and false negative rates | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Salani Mota, Recruiting, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided